CLINICAL TRIAL: NCT02770170
Title: A Double-blind, Randomised, Placebo-controlled Trial Evaluating the Effect of BI 655064 Administered as Sub-cutaneous Injections, on Renal Response After One Year of Treatment, in Patients With Active Lupus Nephritis
Brief Title: Dose Finding, Efficacy and Safety of BI 655064 in Patients With Active Lupus Nephritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1293.10; 2015-001750-15 (EudraCT Number)
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Results first posted 2021-07-12 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- BI 655064 dose 1 (Experimental)
  Interventions: Drug: BI 655064 dose 1
- BI 655064 dose 2 (Experimental)
  Interventions: Drug: BI 655064 dose 2
- BI 655064 dose 3 (Experimental)
  Interventions: Drug: BI 655064 dose 3
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 655064 dose 1
  Arms: BI 655064 dose 1
Drug: BI 655064 dose 2
  Arms: BI 655064 dose 2
Drug: BI 655064 dose 3
  Arms: BI 655064 dose 3
Drug: Placebo
  Arms: Placebo

SUMMARY:
The overall purpose of the study is to assess the efficacy of three different doses of BI 655064 against placebo as add-on therapy to standard of care (SOC) treatment for active lupus nephritis in order to characterize the dose-response relationship within the therapeutic range, and select the target dose for phase III development.

ELIGIBILITY:
Inclusion criteria:

* Males and females 18-70 years. Women of childbearing potential must be ready and able (as assessed by investigator) to use simultaneously two reliable methods of birth control, one of which must be highly effective. Highly effective method, per ICH M3(R2) is a method that result in a low failure rate of less than 1% per year when used consistently and correctly.
* Diagnosis of systemic lupus erythematosus (SLE) by American College of Rheumatology (ACR) criteria 1997, at least 4 criteria must be documented, one of which must be a positive anti-dsDNA antibody OR a positive antinuclear antibody (ANA) at screening or around time of start of induction therapy
* Lupus Nephritis Class III or IV (International Society of Nephrology (ISN)/Renal Pathology Society (RPS) -2003 classification) with either active or active/chronic disease, co-existing class V permitted, proven by renal biopsy within 3 months prior to screening or during screening if induction therapy has not yet been started
* Active renal disease evidenced by proteinuria ≥ 1.0 g/day [(Uprot/Ucrea) ≥ 1]
* Signed and dated written informed consent

Exclusion criteria:

* Clinically significant current other renal disease
* Glomerular Filtration Rate <30ml/min/1.73m²
* Dialysis within 12m of screening
* Antiphospholipid syndrome
* Diabetes mellitus poorly controlled or known diabetic retinopathy or nephropathy
* Evidence of current or previous clinically significant disease, medical condition or finding in the medical examination that in the investigator's opinion would compromise the safety of the patient or the quality of the data
* Any induction therapy for Lupus Nephritis within the last 6 months prior to randomisation except induction with Mycophenolate Mofetil and high dose steroids started within 6 weeks prior to randomisation

  * Treatment with any biologic B-cell depleting therapy (e.g. anti-CD20, anti-CD22,) within 12 months prior to randomisation
  * Treatment with abatacept within 12 months prior to randomisation
  * Treatment with tacrolimus or cyclosporin within 4 weeks prior to randomisation
  * Treatment with cyclophosphamid within 6 months prior to randomisation
  * Treatment with investigational drug within 6 months or 5 half-lives, whichever is greater before randomisation
* Contraindication for MMF or corticosteroids and/or known hypersensitivity to any constituents of the study drug.
* Chronic or relevant acute infections, including but not limited to HIV, Hepatitis B and C and tuberculosis (including a history of clinical tuberculosis (TB) and/or a positive QuantiFERON TB-Gold test
* Any active or suspected malignancy or history of documented malignancy within the last 5 years before screening, except appropriately treated carcinoma in situ and treated basal cell carcinoma.
* Live vaccination within 6 weeks before randomisation
* Patients unable to comply with the protocol in the investigator's opinion.
* Alcohol abuse in the opinion of the investigator or active drug abuse .
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Impaired hepatic function, defined as serum Aspartate Transferase/Alanine Transferase, bilirubin or alkaline phosphatase levels > 2 x Upper Limit of Normal
* Further exclusion criteria apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (74):
- United States (9):
  - Academic Medical Research Institute, Los Angeles, California
  - Integrity Clinical Research, LLC, Doral, Florida
  - Hope Clinical Research, Kissimmee, Florida
  - Integral Rheumatology and Immunology Specialist, Plantation, Florida
  - Emory University, Atlanta, Georgia
  - Northwell Health, Great Neck, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - Office of Dr. Ramesh C. Gupta, Memphis, Tennessee
- Australia (2):
  - The Prince of Wales Hospital, Randwick, New South Wales
  - Princess Alexandra Hospital, Woolloongabba
- Canada (2):
  - Toronto Western Hospital, Toronto, Ontario
  - CHU de Quebec-Universite Laval Research Centre, Québec
- Czechia (3):
  - Hospital Hradec Kralove, Hradec Králové
  - General University Hospital Prague 2, Nephrology Clinic, Prague
  - Institute of Rheumathology Prague, Prague
- France (2):
  - HOP Henri Mondor, Créteil
  - HOP La Pitié Salpêtrière, Paris
- Germany (6):
  - Universitätsklinikum Köln (AöR), Cologne
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart
- Greece (3):
  - General Hospital of Athens "Laiko", Athens
  - University General Hospital Attikon, Athens
  - University General Hospital of Heraklion, Heraklion, Crete
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Azienda Ospedaliera Universitaria di Padova, Padua, Italy
- Japan (7):
  - Hospital of the University of Occupational and Environmental Health, Fukuoka, Kitakyushu
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - St. Marianna University School of Medicine Hospital, Kanagawa, Kawasaki
  - Tohoku University Hospital, Miyagi, Sendai
  - Okayama University Hospital, Okayama, Okayama
  - Juntendo University Hospital, Tokyo, Bunkyo-ku
  - Keio University Hospital, Tokyo, Shinjuku-ku
- Malaysia (2):
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Tengku Ampuan Rahimah, Klang
- Mexico (4):
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - Instituto Nacional de Cs Médicas y Nutrición S Zubiran, Mexico City
  - H. Central Dr Ignacio M. P., San Luis Potosí City
- Philippines (5):
  - Angeles University Foundation Medical Center, Angeles City
  - Chong Hua Hospital, Cebu City
  - Cebu Doctors Hospital, Cebu City, Cebu
  - Southern Philippines Medical Center, Davao City
  - Mary Mediatrix Medical Center, Lipa City, Batangas
- Poland (6):
  - University Clinical Hospital in Bialystok I, Bialystok
  - Norbert Barlicki University Clinical Hospital No.1, Lodz, Lodz
  - Cent.Clin.Hosp.Med.Univ.Lodz,Electrocard, Lodz
  - Clinic Medical Center; Nowa Sol, Nowa Sól
  - NZOZ Centrum Medyczne AESKULAP,Private Prac, Radom, Radom
  - John Paul II Regional Hospital, Zamosc, Zamość
- Portugal (4):
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Hospital Curry Cabral, EPE, Lisbon
  - CHULN, EPE - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar Universitário São João,EPE, Porto
- Serbia (3):
  - Institute of Rheumatology, Belgrade, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Centre Nis, Niš
- Ajou University Hospital, Suwon, South Korea
- Spain (4):
  - Hospital Vall d'Hebron, Barcelona
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Dr. Peset, Valencia
- Thailand (5):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Pramongkutklao Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiangmai University, Chiang Mai
  - Naresuan University Hospital, Muang
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge
  - Leicester General Hospital, Leicester
  - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Jayne DR, Steffgen J, Romero-Diaz J, Bajema I, Boumpas DT, Noppakun K, Amano H, Gomez HM, Satirapoj B, Avihingsanon Y, Chawanasuntorapoj R, Madero M, Naumnik B, Recto R, Fagan N, Revollo I, Wu J, Visvanathan S, Furie R. Clinical and Biomarker Responses to BI 655064, an Antagonistic Anti-CD40 Antibody, in Patients With Active Lupus Nephritis: A Randomized, Double-Blind, Placebo-Controlled, Phase II Trial. Arthritis Rheumatol. 2023 Nov;75(11):1983-1993. doi: 10.1002/art.42557. Epub 2023 Aug 17. PMID 37192040
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a double-blind, randomised, placebo-controlled trial evaluating the effect of BI 655064 administered as subcutaneous injections, on renal response after one year of treatment, in patients with active lupus nephritis.
Pre-assignment Details: All patients were screened for eligibility prior to participation in the trial. Patients attended a specialist site which ensured that they (the patients) strictly met all inclusion and none of the exclusion criteria. Patients were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 120 mg BI 655064: Participants in dose group 1 received two subcutaneous injections per week, one of 120 milligrams (mg) of BI 655064 and one of matching placebo on the same day for 3 weeks followed by one subcutaneous injection per week of 120 mg of BI 655064 alternating with placebo, up to 52 weeks.
- 180 mg BI 655064: Participants in dose group 2 received two subcutaneous injections per week, one of 180 milligrams (mg) of BI 655064 and one of matching placebo on the same day for 3 weeks followed by one subcutaneous injection per week of 180 mg of BI 655064 alternating with placebo, up to 52 weeks.
- 240 mg BI 655064: Participants in dose group 3 received two subcutaneous injections per week of 120 milligrams (mg) of BI 655064 (240 mg in total) on the same day for 3 weeks followed by one subcutaneous injection per week of 120 mg of BI 655064, up to 52 weeks.
- Placebo: Participants in the placebo group received two subcutaneous injections per week of placebo on the same day for 3 weeks followed by one subcutaneous injection per week of placebo, up to 52 weeks.
Period: Overall Study
Arm/Group | 120 mg BI 655064 | 180 mg BI 655064 | 240 mg BI 655064 | Placebo
Started | 21 | 20 | 40 | 40
Completed | 14 | 17 | 35 | 33
Not Completed | 7 | 3 | 5 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — due to pregnancy | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 1
Not completed — Adverse Event | 4 | 3 | 5 | 3
Not completed — due to disease worsening | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set included all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 120 mg BI 655064 | 180 mg BI 655064 | 240 mg BI 655064 | Placebo | Total
Number analyzed (Participants) | 21 | 20 | 40 | 40 | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.9 (11.4) | 34.5 (9.9) | 34.3 (10.3) | 33.9 (9.8) | 34.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 36 | 38 | 108
  Male | 5 | 2 | 4 | 2 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 8 | 7 | 24
  Not Hispanic or Latino | 16 | 16 | 32 | 33 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 9 | 17 | 17 | 52
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 1 | 4
  White | 9 | 11 | 21 | 22 | 63
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
estimated glomerular filtration rate (eGFR) at baseline [Mean (Standard Deviation); unit: mL/min/1.73 m²] — estimated glomerular filtration rate (eGFR) was calculated from serum creatinine.
  mL/min/1.73 m² | 85.857 (34.268) | 99.850 (21.109) | 91.125 (32.673) | 88.775 (29.914) | 90.876 (30.387)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Renal Response (CRR) at Week 52
Description: Complete renal response (CRR) was defined as urine protein (UP) < 0.5 g/day at Week 52 and either estimated glomerular filtration rate (eGFR) within normal range at Week 52 or decrease in eGFR < 20% from baseline at Week 52 if eGFR was below normal range (below lower limit of normal [LLN], where LLN = 90 mL/min).
  CRR at Week 52 (derived using UP from the 24 h urine collections) was analyzed using a logistic regression model. Factors in the model included treatment and the covariates race (Asian/Non-Asian) and proteinuria at screening (UP/urine creatinine (UC) <3 or >=3 g/day).
  Pairwise comparisons of the modelled proportions of patients with CRR at each dose level to placebo were performed.
Time Frame: At week 52.
Population: Intent to treat (ITT) set: This patient set included all patients from the treated set who had a baseline (or screening) proteinuria (spot urine could be used if a patient did not have 24 h urine collections) and a baseline or screening estimated glomerular filtration rate (eGFR) value.
Measure: Number; unit: Percentage of Participants
Arm/Group | 120 mg BI 655064 | 180 mg BI 655064 | 240 mg BI 655064 | Placebo
Number analyzed (Participants) | 21 | 20 | 40 | 40
Percentage of Participants | 38.32 | 44.95 | 44.56 | 48.33
Statistical Analysis 1: Comparison: 120 mg BI 655064 vs 180 mg BI 655064 vs 240 mg BI 655064 vs Placebo; Multiple comparison procedures and modelling (MCPmod) techniques for logistic regression was used; Test type: Other; p = 0.7271, MCPMod quadratic model fit — An alpha of 0.20 was used for one-sided test. The MCPMod procedure adjusts for multiplicity
Statistical Analysis 2: Comparison: 120 mg BI 655064 vs 180 mg BI 655064 vs 240 mg BI 655064 vs Placebo; Multiple comparison procedures and modelling (MCPmod) techniques for logistic regression was used; Test type: Other; p = 0.6415, MCPMod sigmoidal Emax model fit — An alpha of 0.20 was used for one-sided test. The MCPMod procedure adjusts for multiplicity
Statistical Analysis 3: Comparison: 120 mg BI 655064 vs 180 mg BI 655064 vs 240 mg BI 655064 vs Placebo; Multiple comparison procedures and modelling (MCPmod) techniques for logistic regression was used; Test type: Other; p = 0.7367, MCPMod Emax model fit — An alpha of 0.20 was used for one-sided test. The MCPMod procedure adjusts for multiplicity
Statistical Analysis 4: Comparison: 120 mg BI 655064 vs 180 mg BI 655064 vs 240 mg BI 655064 vs Placebo; Multiple comparison procedures and modelling (MCPmod) techniques for logistic regression was used; Test type: Other; p = 0.6624, MCPMod exponential model fit — An alpha of 0.20 was used for one-sided test. The MCPMod procedure adjusts for multiplicity
Statistical Analysis 5: Comparison: 120 mg BI 655064 vs Placebo; Test type: Other; p = 0.4645, Regression, Logistic; include treatment and covariates, race (Asian or non-Asian), proteinuria at screening (<3g/day or >= 3g/day); Risk Difference (RD) = -10.00, 80% CI 2-sided [-27.292 to 7.288] — Confidence intervals calculated using delta method
Statistical Analysis 6: Comparison: 180 mg BI 655064 vs Placebo; Test type: Other; p = 0.8084, Regression, Logistic; include treatment and covariates, race (Asian or non-Asian), proteinuria at screening (<3g/day or >= 3g/day); Risk Difference (RD) = -3.38, 80% CI 2-sided [-21.204 to 14.451] — Confidence intervals calculated using delta method
Statistical Analysis 7: Comparison: 240 mg BI 655064 vs Placebo; Test type: Other; p = 0.7398, Regression, Logistic; include treatment and covariates, race (Asian or non-Asian), proteinuria at screening (<3g/day or >= 3g/day); Risk Difference (RD) = -3.77, 80% CI 2-sided [-18.364 to 10.832] — Confidence intervals calculated using delta method

2. Secondary Outcome: Percentage of Patients With Complete Renal Response (CRR) at Week 26
Description: Complete renal response (CRR) was defined as urine protein (UP) < 0.5 g/day at Week 26 and either estimated glomerular filtration rate (eGFR) within normal range at Week 26 or decrease in eGFR < 20% from baseline at Week 26 if eGFR was below normal range (below lower limit of normal [LLN], where LLN = 90 mL/min).
Time Frame: At week 26.
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 120 mg BI 655064 | 180 mg BI 655064 | 240 mg BI 655064 | Placebo
Number analyzed (Participants) | 21 | 20 | 40 | 40
Percentage of Participants | 28.6 | 50.0 | 35.0 | 37.5
Statistical Analysis 1: Comparison: 120 mg BI 655064 vs Placebo; Test type: Other; p = 0.5773, Barnard test of association; Risk Difference (RD) = -8.93, 80% CI 2-sided [-23.66 to 7.64] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method
Statistical Analysis 2: Comparison: 180 mg BI 655064 vs Placebo; Test type: Other; p = 0.4013, Barnard test of association; Risk Difference (RD) = 12.50, 80% CI 2-sided [-4.59 to 29.03] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method
Statistical Analysis 3: Comparison: 240 mg BI 655064 vs Placebo; Test type: Other; p = 0.8965, Barnard test of association; Risk Difference (RD) = -2.50, 80% CI 2-sided [-15.98 to 11.10] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method

3. Secondary Outcome: Percentage of Patients With Partial Renal Response (PRR) at Week 26
Description: Partial renal response (PRR) was defined as at least 50% reduction of proteinuria from baseline if estimated glomerular filtration rate (eGFR) was within normal range at time of assessment or decrease of eGFR <20% from baseline if eGFR was below normal range at time of assessment.
Time Frame: At week 26.
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 120 mg BI 655064 | 180 mg BI 655064 | 240 mg BI 655064 | Placebo
Number analyzed (Participants) | 21 | 20 | 40 | 40
Percentage of Participants | 42.9 | 75.0 | 62.5 | 62.5
Statistical Analysis 1: Comparison: 120 mg BI 655064 vs Placebo; Test type: Other; p = 0.1476, Barnard test of association; Risk Difference (RD) = -19.64, 80% CI 2-sided [-35.38 to -2.48] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method
Statistical Analysis 2: Comparison: 180 mg BI 655064 vs Placebo; Test type: Other; p = 0.4013, Barnard test of association; Risk Difference (RD) = 12.50, 80% CI 2-sided [-4.20 to 26.86] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method
Statistical Analysis 3: Comparison: 240 mg BI 655064 vs Placebo; Test type: Other; Barnard test of association; Risk Difference (RD) = 0.00, 80% CI 2-sided [-13.63 to 13.63] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method

4. Secondary Outcome: Percentage of Patients With Partial Renal Response (PRR) at Week 52
Description: as for outcome 3
Time Frame: At week 52.
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 120 mg BI 655064 | 180 mg BI 655064 | 240 mg BI 655064 | Placebo
Number analyzed (Participants) | 21 | 20 | 40 | 40
Percentage of Participants | 33.3 | 65.0 | 55.0 | 60.0
Statistical Analysis 1: Comparison: 120 mg BI 655064 vs Placebo; Test type: Other; p = 0.0512, Barnard test of association; Risk Difference (RD) = -26.67, 80% CI 2-sided [-41.52 to -9.42] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method
Statistical Analysis 2: Comparison: 180 mg BI 655064 vs Placebo; Test type: Other; p = 0.7597, Barnard test of association; Risk Difference (RD) = 5.00, 80% CI 2-sided [-12.10 to 20.74] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method
Statistical Analysis 3: Comparison: 240 mg BI 655064 vs Placebo; Test type: Other; p = 0.7505, Barnard test of association; Risk Difference (RD) = -5.00, 80% CI 2-sided [-18.74 to 9.02] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method

5. Secondary Outcome: Percentage of Patients With Major Renal Response (MRR) at Week 26
Description: Major renal response was defined as follows depending on proteinuria at baseline:
  * If baseline proteinuria was <3 g/day and patient had complete renal response (CRR)
  * If baseline proteinuria was >= 3 g/day and proteinuria < 1 g/day and either estimated glomerular filtration rate (eGFR) within normal range or decrease in eGFR <20% from baseline at Week 26 if eGFR was below normal range (below lower limit of normal (LLN), where LLN = 90 mL/min)
Time Frame: At week 26.
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 120 mg BI 655064 | 180 mg BI 655064 | 240 mg BI 655064 | Placebo
Number analyzed (Participants) | 21 | 20 | 40 | 40
Percentage of Participants | 28.6 | 55.0 | 37.5 | 50.0
Statistical Analysis 1: Comparison: 120 mg BI 655064 vs Placebo; Test type: Other; p = 0.1269, Barnard test of association; Risk Difference (RD) = -21.43, 80% CI 2-sided [-36.03 to -4.41] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method
Statistical Analysis 2: Comparison: 180 mg BI 655064 vs Placebo; Test type: Other; p = 0.7889, Barnard test of association; Risk Difference (RD) = 5.00, 80% CI 2-sided [-12.24 to 21.62] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method
Statistical Analysis 3: Comparison: 240 mg BI 655064 vs Placebo; Test type: Other; p = 0.2906, Barnard test of association; Risk Difference (RD) = -12.50, 80% CI 2-sided [-25.99 to 1.68] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method

6. Secondary Outcome: Percentage of Patients With Major Renal Response (MRR) at Week 52
Description: Major renal response was defined as follows depending on proteinuria at baseline:
  * If baseline proteinuria was <3 g/day and patient had complete renal response (CRR)
  * If baseline proteinuria was >= 3 g/day and proteinuria < 1 g/day and either estimated glomerular filtration rate (eGFR) within normal range or decrease in eGFR <20% from baseline at Week 52 if eGFR was below normal range (below lower limit of normal (LLN), where LLN = 90 mL/min)
Time Frame: At week 52.
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 120 mg BI 655064 | 180 mg BI 655064 | 240 mg BI 655064 | Placebo
Number analyzed (Participants) | 21 | 20 | 40 | 40
Percentage of Participants | 42.9 | 55.0 | 52.5 | 52.5
Statistical Analysis 1: Comparison: 120 mg BI 655064 vs Placebo; Test type: Other; p = 0.5687, Barnard test of association; Risk Difference (RD) = -9.64, 80% CI 2-sided [-25.79 to 7.45] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method
Statistical Analysis 2: Comparison: 180 mg BI 655064 vs Placebo; Test type: Other; p = 0.9217, Barnard test of association; Risk Difference (RD) = 2.50, 80% CI 2-sided [-14.67 to 19.17] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method
Statistical Analysis 3: Comparison: 240 mg BI 655064 vs Placebo; Test type: Other; Barnard test of association; Risk Difference (RD) = 0.00, 80% CI 2-sided [-14.03 to 14.03] — Unadjusted absolute risk difference; Confidence intervals calculated using Newcombe method

ADVERSE EVENTS:
Time Frame: From the first does of study medication until end of the 52-week treatment + 8 weeks of follow-up, up to 60 weeks.
Description: Treated set (TS): This patient set included all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Arm/Group | 120 mg BI 655064 | 180 mg BI 655064 | 240 mg BI 655064 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 1/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 6/21 | 6/20 | 10/40 | 8/40
Other Adverse Events (participants affected / at risk) | 17/21 | 13/20 | 34/40 | 35/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 120 mg BI 655064 (N=21) | 180 mg BI 655064 (N=20) | 240 mg BI 655064 (N=40) | Placebo (N=40)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Chorioretinopathy (Eye disorders) | 1 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Genital herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 0 | 0 | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Lupus nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 120 mg BI 655064 (N=21) | 180 mg BI 655064 (N=20) | 240 mg BI 655064 (N=40) | Placebo (N=40)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 4 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 6 | 1
Cushingoid (Endocrine disorders) | 1 | 3 | 2 | 2
Dry eye (Eye disorders) | 0 | 0 | 1 | 3
Vision blurred (Eye disorders) | 2 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 9 | 6
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 3
Asthenia (General disorders) | 2 | 0 | 1 | 1
Fatigue (General disorders) | 2 | 1 | 1 | 1
Injection site pain (General disorders) | 2 | 1 | 3 | 0
Oedema peripheral (General disorders) | 3 | 1 | 3 | 2
Pyrexia (General disorders) | 3 | 0 | 2 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 3
Gastroenteritis (Infections and infestations) | 0 | 1 | 3 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 4 | 3
Nasopharyngitis (Infections and infestations) | 2 | 1 | 4 | 7
Oral candidiasis (Infections and infestations) | 2 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 3
Rhinitis (Infections and infestations) | 0 | 0 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 6 | 7 | 8
Urinary tract infection (Infections and infestations) | 1 | 2 | 4 | 6
Lymphocyte count decreased (Investigations) | 0 | 0 | 3 | 0
Weight increased (Investigations) | 2 | 2 | 5 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 3
Headache (Nervous system disorders) | 3 | 1 | 6 | 5
Insomnia (Psychiatric disorders) | 1 | 2 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 9 | 7
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 6 | 2
Hypertension (Vascular disorders) | 1 | 1 | 2 | 3
Hypotension (Vascular disorders) | 0 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT02770170/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT02770170/SAP_001.pdf